CLINICAL TRIAL: NCT01419223
Title: Patient Beliefs and Attitudes That Influence Participation in PTSD-TBI Clinical Trials
Brief Title: Patient Participation Beliefs and Post-Traumatic Stress Disorder (PTSD)
Status: Completed | Type: Observational
Sponsor: INTRuST, Post-Traumatic Stress Disorder - Traumatic Brain Injury Clinical Consortium (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: INTRuST- Beliefs and Attitudes
Record Dates: First submitted 2011-08-16; First posted 2011-08-18 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Post-Traumatic Stress Disorder; Brain Injuries, Traumatic
Keywords: Qualitative research; Health Knowledge, Attitudes, Practice; Refusal to Participate
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic; Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Consent to participate (Group 1): Active military and veterans who consent to participate in an INTRuST PTSD or TBI research trial.
- Decline to participate (Group 2): Active military and veterans who decline to participate in an INTRuST PTSD or TBI research trial.

SUMMARY:
This is an exploratory qualitative interview study being conducted with a primary objective of examining perceptions held by active military and veterans regarding help-seeking attitudes and mental health beliefs which influence the decision to consent or decline participation in Post-Traumatic Stress Disorder (PTSD) or Traumatic Brain Injury (TBI) clinical trials. Active duty military and/or veterans aged 18 years and older who consent to participate (N = 50), or have recently declined participation (N = 50), in an INTRuST affiliated outpatient clinical trial for deployment-related PTSD or TBI will be recruited. Participants who consent to participate in an INTRuST clinical trial (Group 1) will be interviewed once at the beginning the of the clinical trial, and again following participation in the trial. Participants who decline participation in an INTRuST affiliated outpatient clinical trial (Group 2) will be interviewed once. For participants in both groups, study participation will initiate within 1 month of referral to study. Total duration of study participation is based on the specific clinical trial that the participant is recruitment from; the longest trial is estimated to be 24 weeks or less. Semi-structured qualitative individual interviews will be conducted to carry out a thematic analysis of the data exploring familial, social and institution-level constructs which may influence the subjective experience of the research treatment process.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and over
2. Active duty and/or veteran
3. Referred to participate in INTRuST-affiliated outpatient clinical trials for PTSD or TBI
4. Ability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Active military and/or veterans ages 18 or over who have recently considered participating in an outpatient clinical trial for PTSD or TBI.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Perceptions about participation in clinical trials for PTSD or TBI as measured via qualitative interview. | Qualitative interviews will be conducted during an expected average time frame of 12-24 weeks per study participant based on the specific study recruited from.
  Perceptions regarding help-seeking attitudes and mental health beliefs which influence the decision to consent or decline participation in clinical treatment trials for PTSD-TBI will be measured via serial qualitative interview framework.

SECONDARY OUTCOMES:
Feasibility of conducting qualitative interviews with active duty military and veterans who consent or decline participation in a PTSD or TBI clinical trial as measured by study participation. | End of 21-month study recruitment period
  Feasibility will be determined by the number of participants anticipated vs. the number actually enrolled in the current study.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Hurst, Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States